CLINICAL TRIAL: NCT04015544
Title: Expression of Systemic Markers of Atherosclerosis in Free-living, Overweight, Postmenopausal Women Following Daily Watermelon Consumption for Six Weeks: A Randomized Controlled Trial
Brief Title: Markers of Atherosclerosis in Overweight, Postmenopausal Women Following Daily Watermelon Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: National Watermelon Promotion Board; https://www.watermelon.org (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14-0092
Record Dates: First submitted 2019-07-02; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Postmenopausal; Overweight and Obesity
Keywords: insulin; glucose; cardiovascular disease; inflammation; watermelon; L-citrulline; L-arginine
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watermelon (Experimental): Watermelon puree 710 mL per day for six weeks
  Interventions: Dietary Supplement: Watermelon
- Control (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Watermelon — Pureed whole (100%) watermelon
  Arms: Watermelon

SUMMARY:
The primary purpose of this study is to determine the effectiveness of six weeks of watermelon puree supplementation, compared to control (no treatment), on blood antioxidant capacity, inflammation markers in the blood, biomarkers of metabolism in the blood, and cardiovascular disease markers in the blood, and biomarkers in the blood related to watermelon ingestion in overweight post-menopausal women. The secondary purpose is to compare body composition and body mass between the watermelon supplement group and the control group.

DETAILED DESCRIPTION:
ORIENTATION AND PRE-STUDY TESTING (1-2 hours):

1. Come to the Lab in the morning in an overnight fasted state.
2. Complete orientation to the study, and provide voluntary consent to join the study.
3. Complete a medical health questionnaire to verify medical history and lifestyle habits, and provide a 3-day food record.
4. Record symptoms on a questionnaire regarding how subjects have felt for the previous four weeks using a 12-point Likert scale. Symptoms relate to digestive health, hunger, energy, infection, pain, allergies, stress, mental focus, and overall wellbeing.
5. All forms reviewed to determine eligibility to participate in this study.
6. Subject height, body weight, and percent body fat measured.
7. A blood sample taken by a trained phlebotomist; the sample not to exceed 40 mL. Blood tested for markers associated with inflammation and cardiovascular health, and nutritional compounds related to drinking watermelon puree.
8. Subjects randomized to the Control or Watermelon group. If assigned to the Watermelon group subjects provided a six-week supply of watermelon puree.
9. The morning of the study subjects consume the three bottles of watermelon puree (710 mL total, Watermelon group) each day thereafter for six weeks or maintain normal daily fluid intake (Control group).
10. Six weeks after beginning the study subjects return to the Laboratory for the final measurements. Subjects to bring all beverage bottles.

6-WEEK LAB VISIT (1-2 hours):

1. Participants come to the Lab in the morning in an overnight fasted state.
2. Subject body weight, and percent body fat are measured.
3. Subjects record symptoms on a questionnaire regarding how they have felt for the previous six weeks.
4. A final blood sample (40 mL) taken by a trained phlebotomist.

BLOOD SAMPLE ANALYSES

1. Blood borne cardiovascular disease markers: ADAM metallopeptidase with thrombospondin type 1 motif, 13 (ADAMTS13), soluble vascular cell adhesion molecule-1 (sVCAM-1), soluble P-selectin (sP-selectin), growth differentiation factor-15 (GDF-15), and soluble intercellular adhesion molecule-1 (sICAM-1) measured according to the manufacturer's specifications using the MAGPIX instrument and xPONENT analysis software (Luminex, Austin, TX).
2. Fasting blood glucose, insulin, vitamin C, and high-sensitivity C-reactive (hs-CRP) protein were measured by LabCorp (Burlington, NC).
3. Fasting plasma carotenoid concentrations measured commercially (Craft Technologies Inc., Wilson, NC).
4. Fasting plasma amino acid concentration determined by high-performance liquid chromatography.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 50 to 75 years of age,
* have not menstruated for at least 1 year (menopause),
* have a BMI of ≥25 kg/m2,
* nonsmoker with
* no diagnosed history of chronic diseases including: coronary heart disease, stroke, cancer, type 1 or 2 diabetes mellitus, or rheumatoid arthritis;
* may not regularly consume large quantities of L-citrulline/L-arginine rich foods (red meat, tuna fish, cheese, nuts),
* may not regularly take L-citrulline/L-arginine supplements,
* may not use anti-hypertension medications (including diuretic medications),
* may not use exogenous ovarian hormones, or
* may not use medications known to influence inflammation within the two weeks of the study period (specifically non-steroidal anti-inflammatory drugs; NSAIDS).

Exclusion Criteria:

* Male,
* younger than 50 or older than 75 years of age,
* menstruated within the last year,
* have a BMI of <25 kg/m2, smoker,
* diagnosed history of chronic diseases including: coronary heart disease, stroke, cancer, type 1 or 2 diabetes mellitus, or rheumatoid arthritis;
* regularly consume large quantities of L-citrulline/L-arginine rich foods (red meat, tuna fish, cheese, nuts),
* regularly take L-citrulline/L-arginine supplements,
* use anti-hypertension medications (including diuretic medications),
* use exogenous ovarian hormones, or
* use medications known to influence inflammation within the two weeks of the study period (specifically non-steroidal anti-inflammatory drugs; NSAIDS).

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in select plasma cardiovascular disease markers | Pre-study and study completion (6 weeks)
  Plasma concentrations of ADAMTS13, sVCAM-1, sP-selectin, GDF-15, hs-CRP, and sICAM-1

SECONDARY OUTCOMES:
Blood glucose | Pre-study and study completion (6 weeks)
  Fasting blood glucose
Blood insulin | Pre-study and study completion (6 weeks)
  Fasting blood insulin
Blood carotenoids | Pre-study and study completion (6 weeks)
  Fasting blood carotenoids
Blood amino acids | Pre-study and study completion (6 weeks)
  Fasting blood amino acids
Body mass | Pre-study and study completion (6 weeks)
  Body mass (kg)
Body mass index | Pre-study and study completion (6 weeks)
  Body mass index (kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: R. Andrew Shanely, Ph.D., Principal Investigator — Appalachian State University
Locations (1):
- Appalachian State University, Boone, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collins JK, Wu G, Perkins-Veazie P, Spears K, Claypool PL, Baker RA, Clevidence BA. Watermelon consumption increases plasma arginine concentrations in adults. Nutrition. 2007 Mar;23(3):261-6. doi: 10.1016/j.nut.2007.01.005. PMID 17352962
- [Background] Kannel WB, Hjortland MC, McNamara PM, Gordon T. Menopause and risk of cardiovascular disease: the Framingham study. Ann Intern Med. 1976 Oct;85(4):447-52. doi: 10.7326/0003-4819-85-4-447. PMID 970770
- [Background] Lum T, Connolly M, Marx A, Beidler J, Hooshmand S, Kern M, Liu C, Hong MY. Effects of Fresh Watermelon Consumption on the Acute Satiety Response and Cardiometabolic Risk Factors in Overweight and Obese Adults. Nutrients. 2019 Mar 12;11(3):595. doi: 10.3390/nu11030595. PMID 30870970
- [Background] Edwards AJ, Vinyard BT, Wiley ER, Brown ED, Collins JK, Perkins-Veazie P, Baker RA, Clevidence BA. Consumption of watermelon juice increases plasma concentrations of lycopene and beta-carotene in humans. J Nutr. 2003 Apr;133(4):1043-50. doi: 10.1093/jn/133.4.1043. PMID 12672916
- [Background] Cook-Mills JM, Marchese ME, Abdala-Valencia H. Vascular cell adhesion molecule-1 expression and signaling during disease: regulation by reactive oxygen species and antioxidants. Antioxid Redox Signal. 2011 Sep 15;15(6):1607-38. doi: 10.1089/ars.2010.3522. Epub 2011 May 11. PMID 21050132